CLINICAL TRIAL: NCT03659955
Title: Autologous Blood in the Treatment of Severe Dry Eyes and Ocular Surface Disease
Brief Title: Autologous Blood Treatment for Ocular Surface Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lanarkshire (Other Government)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); NHS Research Scotland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L17047
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Ocular Surface Disease
Keywords: Dry eye; Ocular surface; Autologous blood
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Cross sectional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous blood (Experimental): Patients with severe dry eye and ocular surface disease who attend the corneal service within NHS Lanarkshire and who are unresponsive to conservative treatment measures will be considered for treatment of their condition with autologous blood.
  Intervention is application of autologous blood.
  Interventions: Other: Autologous blood applied to dry eye

INTERVENTIONS:
Other: Autologous blood applied to dry eye — See previous description for the study arm.

SUMMARY:
In this study, we aim to determine the efficacy of autologous blood as an alternative to autologous serum eye drops (ASE) in people with severe dry eyes and ocular surface inflammation. ASE are drops manufactured from the patient's own blood. Perceived benefits are that human blood contains multiple components that are beneficial to healing and maintaining a healthy ocular surface, including epidermal growth factor, and transforming growth factor β, in addition to fibronectin, vitamin A, and various growth factors. We wish to assess whether administering autologous blood directly to their eye would also be an effective treatment in the management of severe dry eye. It will be the first study analysing the potential benefits of this relatively novel treatment in Scotland and will consider its role in treating an important debilitating condition.

DETAILED DESCRIPTION:
The surface of the eye, including the cornea, is dependent on the tear film to protect it. An adequate tear film prevents epithelial breakdown, ulceration and secondary infection. The continual regeneration of the corneal epithelium is supported by various components that reside in human tears, such as growth factors, vitamins, electrolytes and neuropeptides. There are various ocular conditions that can lead to a deficiency in any of these tear constituents and can result in excessive surface dryness. This can lead to corneal surface breakdown, non-healing ulceration, secondary infection, globe perforation and sight loss, in addition to severe pain for patients, all of which can have a significant negative impact on a patient's quality of life. First line therapy in the treatment of tear deficiency is in the form of ocular lubricants. Multiple formulations are available in drop, gel and ointment form. Lubricants act as barriers in one form or another to protect the epithelial surface from mechanical trauma. However, in the presence of an unhealthy tear film or corneal epithelial surface, barrier protection alone is inadequate to promote surface regeneration and wound healing. Therefore, even the use of frequent and continual ocular lubricants may be of no benefit to patients with severe ocular surface disease (OSD).

In this study, we aim to determine the efficacy of autologous blood as an alternative to autologous serum eye drops (ASE) in people with severe dry eyes and ocular surface inflammation. ASE are drops manufactured from the patient's own blood. Perceived benefits are that human blood contains multiple components that are beneficial to healing and maintaining a healthy ocular surface, including epidermal growth factor, and transforming growth factor β, in addition to fibronectin, vitamin A, and various growth factors. We wish to assess whether administering autologous blood directly to their eye would also be an effective treatment in the management of severe dry eye. It will be the first study analysing the potential benefits of this relatively novel treatment in Scotland and will consider its role in treating an important debilitating condition.

ELIGIBILITY:
Inclusion Criteria:

1. Known dry eye and ocular surface disease with or without persistent epithelial defect.
2. No improvement in clinical condition after minimum of six months treatment with conventional ocular lubricants.
3. No improvement in clinical condition after treatment of all other potential sources of ocular surface disease, including localised and systemic inflammatory disease.
4. All topical treatments for dry eye and any other pre-existing ocular conditions are preservative free.
5. Patient has capacity to consent to participate in study and to be taught how to administer blood sample.
6. Patients aged between 18-100 years.

Exclusion Criteria:

1. Physical disability preventing patient performing needlestick blood sampling.
2. Concurrent ocular infection.
3. Globe perforation.
4. Patients with known blood borne infections.
5. Patients without capacity to consent to participate in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Ocular surface staining score | 12 months
  To evaluate if the use of autologous blood as described in this study will improve the health of the ocular surface as measured by the ocular surface staining score using the Oxford Grading Scheme.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Lyall, FRCOphth, Principal Investigator — NHS Lanarkshire
Locations (1):
- Hairmyres Hospital, East Kilbride, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No